CLINICAL TRIAL: NCT00294723
Title: Liraglutide Effect and Action in Diabetes (LEAD-3): Effect on Glycemic Control of Liraglutide Versus Glimepiride in Type 2 Diabetes
Brief Title: To Evaluate the Effect of Liraglutide Versus Glimepiride (Amaryl®) on Haemoglobin A1c
Acronym: LEAD-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was terminated at week 195 due to an insufficient number of subjects remaining to obtain reasonable statistical power
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1573; NCT00853359 (obsolete NCT alias)
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Results first posted 2010-03-12 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lira 1.8 (Experimental): Liraglutide 1.8 mg once daily + glimepiride placebo 8 mg once daily, weeks 0-52 (double-blinded period) and open-label liraglutide 1.8 mg once daily in the extension periods (weeks 52-195).
  Interventions: Drug: liraglutide; Drug: placebo
- Lira 1.2 (Experimental): Liraglutide 1.2 mg once daily + glimepiride placebo 8 mg once daily, weeks 0-52 (double-blinded period) and open-label liraglutide 1.2 mg once daily in the extension periods (weeks 52-195).
  Interventions: Drug: liraglutide; Drug: placebo
- Glimepiride - 1 (Active Comparator): Glimepiride 8 mg once daily + liraglutide placebo 200 mcl, weeks 0-52 (double-blinded period) and open-label glimepiride 8 mg once daily in the extension periods (weeks 52-195).
  Interventions: Drug: glimepiride; Drug: placebo
- Glimepiride - 2 (Active Comparator): Glimepiride 8 mg once daily + liraglutide placebo 300 mcl, weeks 0-52 (double-blinded period) and open-label glimepiride 8 mg once daily in the extension periods (weeks 52-195).
  Interventions: Drug: glimepiride; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 1.8 mg for s.c. (under the skin) injection
  Arms: Lira 1.8
Drug: glimepiride — 8 mg capsule
  Arms: Glimepiride - 1; Glimepiride - 2
Drug: liraglutide — 1.2 mg for s.c. (under the skin) injection
  Arms: Lira 1.2
Drug: placebo — Glimepiride placebo, 8mg capsule
  Arms: Lira 1.2; Lira 1.8
Drug: placebo — Liraglutide placebo, 200 mcl
  Arms: Glimepiride - 1
Drug: placebo — Liraglutide placebo, 300 mcl
  Arms: Glimepiride - 2

SUMMARY:
This trial is conducted in North America (the United States of America (USA) and Mexico).

The trial is designed to evaluate the effects of treatment with liraglutide versus glimepiride in subjects with type 2 diabetes. The trial is a 52-week randomised, double-blind trial period plus a 52-week open-label extension (week 104) followed by an additional 156-week continued open-label extension. The total duration of the treatment period is planned to be 260 weeks (5 years).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* TTreatment with diet/exercise or with not more than half maximal dose of oral anti-diabetic drugs alone for at least 2 months
* Diet/exercise treated subjects with HbA1c between 7.0% and 11%, inclusive
* OAD (oral anti-diabetic drug) treated subjects with HbA1c between 7.0% and 10%, inclusive
* Body Mass Index (BMI) less than or equal to 45 kg/m^2

Exclusion Criteria:

* Treatment with insulin for the last 3 months, except short-term treatment for intercurrent illness
* Treatment with any drug that could interfere with the glucose level (besides use of a single anti-diabetic compound)
* Any serious medical condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2006-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (99):
- United States (86):
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Inglewood, California
  - Novo Nordisk Investigational Site, Mission Viejo, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Vista, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Daytona Beach, Florida
  - Novo Nordisk Investigational Site, Delray Beach, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Longwood, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Saint Cloud, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Blue Ridge, Georgia
  - Novo Nordisk Investigational Site, Columbus, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Powder Springs, Georgia
  - Novo Nordisk Investigational Site, Tucker, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Maywood, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Shawnee Mission, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Saint Paul, Minnesota
  - Novo Nordisk Investigational Site, Jackson, Mississippi
  - Novo Nordisk Investigational Site, Tupelo, Mississippi
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Reno, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Plainsboro, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Lewiston, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Bend, Oregon
  - Novo Nordisk Investigational Site, Eugene, Oregon
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Lancaster, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, East Providence, Rhode Island
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Edmonds, Washington
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Tacoma, Washington
- Mexico (12):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Cuernavaca, Morelos
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
  - Novo Nordisk Investigational Site, Chihuahua, Chih
  - Novo Nordisk Investigational Site, Ciudad de México, D.F.
  - Novo Nordisk Investigational Site, Guadalajara
  - Novo Nordisk Investigational Site, Hermosillo, Son.
  - Novo Nordisk Investigational Site, Mexico City
  - Novo Nordisk Investigational Site, Monterrey, N.L.
  - Novo Nordisk Investigational Site, Monterrey, NL
  - Novo Nordisk Investigational Site, Santiago de Querétaro, Qro.
  - Novo Nordisk Investigational Site, Tampico
- Novo Nordisk Investigational Site, Rio Piedras, Puerto Rico

REFERENCES:
- [Result] Garber A, Henry R, Ratner R, Garcia-Hernandez PA, Rodriguez-Pattzi H, Olvera-Alvarez I, Hale PM, Zdravkovic M, Bode B; LEAD-3 (Mono) Study Group. Liraglutide versus glimepiride monotherapy for type 2 diabetes (LEAD-3 Mono): a randomised, 52-week, phase III, double-blind, parallel-treatment trial. Lancet. 2009 Feb 7;373(9662):473-81. doi: 10.1016/S0140-6736(08)61246-5. Epub 2008 Sep 24. PMID 18819705
- [Result] Sullivan SD, Alfonso-Cristancho R, Conner C, Hammer M, Blonde L. Long-term outcomes in patients with type 2 diabetes receiving glimepiride combined with liraglutide or rosiglitazone. Cardiovasc Diabetol. 2009 Feb 26;8:12. doi: 10.1186/1475-2840-8-12. PMID 19245711
- [Result] McGill JB. Insights from the Liraglutide Clinical Development Program--the Liraglutide Effect and Action in Diabetes (LEAD) studies. Postgrad Med. 2009 May;121(3):16-25. doi: 10.3810/pgm.2009.05.1998. PMID 19491536
- [Result] Blonde L, Russell-Jones D. The safety and efficacy of liraglutide with or without oral antidiabetic drug therapy in type 2 diabetes: an overview of the LEAD 1-5 studies. Diabetes Obes Metab. 2009 Dec;11 Suppl 3:26-34. doi: 10.1111/j.1463-1326.2009.01075.x. PMID 19878259
- [Result] Jendle J, Nauck MA, Matthews DR, Frid A, Hermansen K, During M, Zdravkovic M, Strauss BJ, Garber AJ; LEAD-2 and LEAD-3 Study Groups. Weight loss with liraglutide, a once-daily human glucagon-like peptide-1 analogue for type 2 diabetes treatment as monotherapy or added to metformin, is primarily as a result of a reduction in fat tissue. Diabetes Obes Metab. 2009 Dec;11(12):1163-72. doi: 10.1111/j.1463-1326.2009.01158.x. PMID 19930006
- [Result] Bode BW, Testa MA, Magwire M, Hale PM, Hammer M, Blonde L, Garber A; LEAD-3 Study Group. Patient-reported outcomes following treatment with the human GLP-1 analogue liraglutide or glimepiride in monotherapy: results from a randomized controlled trial in patients with type 2 diabetes. Diabetes Obes Metab. 2010 Jul;12(7):604-12. doi: 10.1111/j.1463-1326.2010.01196.x. PMID 20590735
- [Result] Buse JB, Garber A, Rosenstock J, Schmidt WE, Brett JH, Videbaek N, Holst J, Nauck M. Liraglutide treatment is associated with a low frequency and magnitude of antibody formation with no apparent impact on glycemic response or increased frequency of adverse events: results from the Liraglutide Effect and Action in Diabetes (LEAD) trials. J Clin Endocrinol Metab. 2011 Jun;96(6):1695-702. doi: 10.1210/jc.2010-2822. Epub 2011 Mar 30. PMID 21450987
- [Result] Bode BW, Brett J, Falahati A, Pratley RE. Comparison of the efficacy and tolerability profile of liraglutide, a once-daily human GLP-1 analog, in patients with type 2 diabetes >/=65 and <65 years of age: a pooled analysis from phase III studies. Am J Geriatr Pharmacother. 2011 Dec;9(6):423-33. doi: 10.1016/j.amjopharm.2011.09.007. Epub 2011 Nov 4. PMID 22055210
- [Result] Henry RR, Buse JB, Sesti G, Davies MJ, Jensen KH, Brett J, Pratley RE. Efficacy of antihyperglycemic therapies and the influence of baseline hemoglobin A(1C): a meta-analysis of the liraglutide development program. Endocr Pract. 2011 Nov-Dec;17(6):906-13. doi: 10.4158/ep.17.6.906. PMID 22193143
- [Result] Ingwersen SH, Khurana M, Madabushi R, Watson E, Jonker DM, Le Thi TD, Jacobsen LV, Tornoe CW. Dosing rationale for liraglutide in type 2 diabetes mellitus: a pharmacometric assessment. J Clin Pharmacol. 2012 Dec;52(12):1815-23. doi: 10.1177/0091270011430504. Epub 2011 Dec 15. PMID 22174428
- [Result] Zinman B, Schmidt WE, Moses A, Lund N, Gough S. Achieving a clinically relevant composite outcome of an HbA1c of <7% without weight gain or hypoglycaemia in type 2 diabetes: a meta-analysis of the liraglutide clinical trial programme. Diabetes Obes Metab. 2012 Jan;14(1):77-82. doi: 10.1111/j.1463-1326.2011.01493.x. Epub 2011 Oct 30. PMID 21883806
- [Result] Niswender K, Pi-Sunyer X, Buse J, Jensen KH, Toft AD, Russell-Jones D, Zinman B. Weight change with liraglutide and comparator therapies: an analysis of seven phase 3 trials from the liraglutide diabetes development programme. Diabetes Obes Metab. 2013 Jan;15(1):42-54. doi: 10.1111/j.1463-1326.2012.01673.x. Epub 2012 Sep 9. PMID 22862847
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] King AB, Montanya E, Pratley RE, Blonde L, Svendsen CB, Donsmark M, Sesti G. Liraglutide achieves A1C targets more often than sitagliptin or exenatide when added to metformin in patients with type 2 diabetes and a baseline A1C <8.0%. Endocr Pract. 2013 Jan-Feb;19(1):64-72. doi: 10.4158/EP12232.OR. PMID 23186975
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- [Result] Gilbert MP, Marre M, Holst JJ, Garber A, Baeres FM, Thomsen H, Pratley RE. COMPARISON OF THE LONG-TERM EFFECTS OF LIRAGLUTIDE AND GLIMEPIRIDE MONOTHERAPY ON BONE MINERAL DENSITY IN PATIENTS WITH TYPE 2 DIABETES. Endocr Pract. 2016 Apr;22(4):406-11. doi: 10.4158/EP15758.OR. Epub 2015 Nov 17. PMID 26574791
- [Result] Davidson JA, Orsted DD, Campos C. Efficacy and safety of liraglutide, a once-daily human glucagon-like peptide-1 analogue, in Latino/Hispanic patients with type 2 diabetes: post hoc analysis of data from four phase III trials. Diabetes Obes Metab. 2016 Jul;18(7):725-8. doi: 10.1111/dom.12653. Epub 2016 Apr 28. PMID 26936426
- [Derived] Fonseca VA, Devries JH, Henry RR, Donsmark M, Thomsen HF, Plutzky J. Reductions in systolic blood pressure with liraglutide in patients with type 2 diabetes: insights from a patient-level pooled analysis of six randomized clinical trials. J Diabetes Complications. 2014 May-Jun;28(3):399-405. doi: 10.1016/j.jdiacomp.2014.01.009. Epub 2014 Jan 21. PMID 24561125
- [Derived] Hegedus L, Moses AC, Zdravkovic M, Le Thi T, Daniels GH. GLP-1 and calcitonin concentration in humans: lack of evidence of calcitonin release from sequential screening in over 5000 subjects with type 2 diabetes or nondiabetic obese subjects treated with the human GLP-1 analog, liraglutide. J Clin Endocrinol Metab. 2011 Mar;96(3):853-60. doi: 10.1210/jc.2010-2318. Epub 2011 Jan 5. PMID 21209033
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 138 centres in two countries: United States of America (USA) (126) and Mexico (12).
Pre-assignment Details: Subjects with type 2 diabetes treated with diet/exercise or OAD (Oral Anti-Diabetic Drug) monotherapy for at least 2 months were eligible. One subject randomised to the liraglutide 1.8 mg group was withdrawn from the study prior to dosing due to protocol non compliance, subject was not included in the intent-to-treat (ITT) or safety analysis sets.
Groups:
- Glimepiride: Glimepiride 8 mg once daily + liraglutide placebo 200 mcl or liraglutide placebo 300 mcl, weeks 0-52 (double-blinded period) and open-label glimepiride 8 mg once daily in the extension periods (weeks 52-195)
Period: Double-Blind Period 52 Weeks
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Started | 247 (Randomised) | 251 (Randomised) | 248 (Randomised)
Exposed to Study Drug | 246 (Subject withdrew before exposure to drug, and thus not included in the safety and ITT analysis sets) | 251 | 248
Completed | 173 | 162 | 152
Not Completed | 74 | 89 | 96
Not completed — Adverse Event | 18 | 25 | 15
Not completed — Lack of Efficacy | 9 | 15 | 25
Not completed — Protocol Violation | 11 | 11 | 5
Not completed — Not specified in study report | 36 | 38 | 51
Period: Open-Label Extension 52 Weeks
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Started | 154 (19 subjects did not continue into the extension period) | 149 (13 subjects did not continue into the extension period) | 137 (15 subjects did not continue into the extension period)
Completed | 114 | 110 | 97
Not Completed | 40 | 39 | 40
Not completed — Adverse Event | 5 | 5 | 2
Not completed — Lack of Efficacy | 12 | 15 | 21
Not completed — Protocol Violation | 4 | 3 | 3
Not completed — Not specified in study report | 19 | 16 | 14
Period: Additional Open-Label Extension 91 Weeks
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Started | 62 (52 subjects did not continue into the extension period) | 53 (57 subjects did not continue into the extension period) | 28 (69 subjects did not continue into the extension period)
Completed | 34 | 32 | 8
Not Completed | 28 | 21 | 20
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lack of Efficacy | 24 | 14 | 16
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Not specified in study report | 2 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride | Total
Number analyzed (Participants) | 247 | 251 | 248 | 746
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 222 | 208 | 208 | 638
  >=65 years | 25 | 43 | 40 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (10.8) | 53.7 (11.0) | 53.4 (10.9) | 53.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 134 | 115 | 375
  Male | 121 | 117 | 133 | 371
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 87 | 81 | 93 | 261
  Not Hispanic or Latino | 160 | 170 | 155 | 485
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 5 | 9 | 26
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 30 | 34 | 30 | 94
  White | 186 | 200 | 192 | 578
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 17 | 12 | 17 | 46
Region of Enrollment [Number; unit: participants]
  Mexico | 52 | 53 | 66 | 171
  United States | 195 | 198 | 182 | 575
Previous anti-diabetic treatment [Number; unit: participants]
  Diet/Exercise | 87 | 91 | 94 | 272
  Monotherapy | 160 | 160 | 154 | 474
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.8 (6.3) | 33.2 (5.6) | 33.2 (5.6) | 33.1 (5.8)
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 5.3 (5.1) | 5.2 (5.5) | 5.6 (5.1) | 5.4 (5.3)
HbA1c (Glycosylated Haemoglobin A1c) [Mean (Standard Deviation); unit: percentage of total haemoglobin] — HbA1c at screening
  percentage of total haemoglobin | 8.3 (1.1) | 8.3 (1.0) | 8.4 (1.2) | 8.3 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c) at Week 52
Description: Percentage point change in Glycosylated Haemoglobin A1c (HbA1c) from baseline (week 0) to 52 weeks (end of double-blind period)
Time Frame: week 0, week 52
Population: Intention to treat (ITT) analysis set using LOCF (Last Observation Carried Forward) is all randomised subjects who had been exposed to at least one dose of the study products.
Measure: Least Squares Mean (Standard Error); unit: percentage point of total HbA1c
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 234 | 236 | 241
percentage point of total HbA1c | -1.14 (0.08) | -0.84 (0.08) | -0.51 (0.08)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in glycosylated haemoglobin (HbA1c) from baseline to end of treatment at 52 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous oral antidiabetic drug (OAD) treatment as fixed effects and baseline HbA1c as covariate; Test type: Non-Inferiority or Equivalence — The two sided 95% confidence interval for the treatment difference [liraglutide - glimepiride] was estimated. Liraglutide was shown to be non-inferior to glimepiride if the upper limit of the two-sided 95% CI for the treatment difference was below 0.4% and superior if the complete confidence interval was below 0%; p < 0.0001, ANCOVA — The statistical analysis of the primary endpoint was done in a hierarchal manner due to multiple comparisons. No other adjustments were made for multiplicity. 2-sided significance level 5%; Estimated treatment difference, LS Mean = -0.62, 95% CI [-0.83 to -0.42]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The two sided 95% confidence interval for the treatment difference [liraglutide - glimepiride] was estimated. Liraglutide was shown to be non-inferior to glimepiride if the upper limit of the two-sided 95% CI for the treatment difference was below 0.4% and superior if the complete confidence interval was below 0%. Superiority of 1.2 mg liraglutide was only tested if 1.2 mg liraglutide was non-inferior to glimepiride and 1.8 mg liraglutide was superior to glimepiride; p = 0.0014, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Estimated treatment difference, LS Mean = -0.33, 95% CI [-0.53 to -0.13]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — A test for superiority of liraglutide 1.8 mg to liraglutide 1.2 mg was performed to compare the two doses. Superiority of liraglutide 1.8 mg was concluded if the upper limit of the 2-sided 95% CI for the treatment difference (liraglutide 1.8 mg - liraglutide 1.2 mg) was below 0%; p = 0.0046, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -0.29, 95% CI [-0.50 to -0.09]

2. Secondary Outcome: Change in Body Weight at Week 52
Description: Change in body weight from baseline (week 0) to 52 weeks (end of double-blind period)
Time Frame: week 0, week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 240 | 245 | 248
kg | -2.45 (0.28) | -2.05 (0.28) | 1.12 (0.27)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in body weight from baseline to end of treatment at 52 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline body weight as covariate; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.8 mg and glimepiride was calculated. If the upper limit of the 95% CI was below 0 kg, it was concluded that the given dose of liraglutide was better than glimepiride; p < .0001, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -3.58, 95% CI [-4.28 to -2.87]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.2 mg and glimepiride was calculated. If the upper limit of the 95% CI was below 0 kg, it was concluded that the given dose of liraglutide was better than glimepiride; p < .0001, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -3.17, 95% CI [-3.87 to -2.47]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.8 mg and liraglutide 1.2 mg was calculated. If the upper limit of the 95% CI was below 0 kg, it was concluded that the liraglutide 1.8 mg was better than liraglutide 1.2 mg; p = 0.2584, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -0.41, 95% CI [-1.11 to 0.30]

3. Secondary Outcome: Change in Body Weight at Week 104
Description: Change in body weight from baseline (week 0) to 104 weeks (end of 52-week extension)
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 240 | 245 | 248
kg | -2.70 (0.32) | -1.89 (0.31) | 0.95 (0.30)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in body weight from baseline to end of treatment at 104 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline body weight as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < .0001, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -3.65, 95% CI [-4.44 to -2.86]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < .0001, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -2.84, 95% CI [-3.63 to -2.06]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p = 0.0462, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -0.80, 95% CI [-1.59 to -0.01]

4. Primary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c) at Week 104
Description: Percentage point change in Glycosylated Haemoglobin A1c (HbA1c) from baseline (week 0) to 104 weeks (end of 52-week extension)
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage point of total HbA1c
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 234 | 236 | 241
percentage point of total HbA1c | -0.88 (0.09) | -0.59 (0.09) | -0.28 (0.09)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in glycosylated haemoglobin (HbA1c) from baseline to end of treatment at 104 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous oral antidiabetic drug (OAD) treatment as fixed effects and baseline HbA1c as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < .0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Estimated treatment difference, LS Mean = -0.60, 95% CI [-0.83 to -0.38]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — The two sided 95% CI for the treatment difference [liraglutide - glimepiride] was estimated. Liraglutide was non-inferior to glimepiride if the upper limit of the two-sided 95% CI for the treatment difference was below 0.4% and superior if the complete confidence interval was below 0%. Superiority of 1.2 mg liraglutide was only tested if 1.2 mg liraglutide was non-inferior to glimepiride and 1.8 mg liraglutide was superior to glimepiride; p = 0.0076, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Estimated treatment difference, LS Mean = -0.31, 95% CI [-0.54 to -0.08]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.0129, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -0.29, 95% CI [-0.52 to -0.06]

5. Secondary Outcome: Change in Body Weight at Week 156
Description: Change in body weight from baseline (week 0) to 156 weeks
Time Frame: week 0, week 156
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 240 | 245 | 248
kg | -2.43 (0.32) | -1.68 (0.32) | 1.05 (0.31)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in body weight from baseline to end of treatment at 156 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country, and previous anti-diabetic treatment as fixed effects and baseline body weight as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA — 2-sided significance level was 5%; Estimated treatment difference, LS Mean = -3.48, 95% CI [-4.28 to -2.68]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.0001, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -2.72, 95% CI [-3.52 to -1.93]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; Change in body weight from baseline to end of treatment at 156 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country, and previous anti-diabetic treatment as fixed effects and baseline body weight as covariance; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p = 0.0642, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -0.75, 95% CI [-1.55 to 0.05]

6. Secondary Outcome: Change in Fasting Plasma Glucose at Week 52
Description: Change in fasting plasma glucose (FPG) from baseline (week 0) to 52 weeks (end of double-blind period)
Time Frame: week 0, week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 230 | 234 | 242
mg/dL | -25.57 (3.50) | -15.21 (3.50) | -5.29 (3.33)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in fasting plasma glucose (FPG) from baseline to end of treatment at 52 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline FPG as covariate; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.8 mg and glimepiride was calculated. If the upper limit of the 95% CI was below 0 mg/dL, it was concluded that the given dose of liraglutide was better than glimepiride; p < .0001, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -20.28, 95% CI [-29.09 to -11.46]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.2 mg and glimepiride was calculated. If the upper limit of the 95% CI was below 0 mg/dL, it was concluded that the given dose of liraglutide was better than glimepiride; p = 0.0270, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -9.92, 95% CI [-18.70 to -1.12]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 6, analysis 1]; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the treatment difference between liraglutide 1.8 mg and liraglutide 1.2 mg was calculated. If the upper limit of the 95% CI was below 0 mg/dL, it was concluded that liraglutide 1.8 mg was better than liraglutide 1.2 mg; p = 0.0223, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -10.36, 95% CI [-19.24 to -1.48]

7. Secondary Outcome: Change in Fasting Plasma Glucose at Week 104
Description: Change in fasting plasma glucose (FPG) from baseline (week 0) to 104 weeks (end of 52-week extension)
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 230 | 234 | 242
mg/dL | -15.82 (3.85) | -9.36 (3.85) | 1.97 (3.66)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in fasting plasma glucose (FPG) from baseline to end of treatment at 104 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline FPG as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.0003, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -17.79, 95% CI [-27.48 to -8.09]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 2]; p = 0.0217, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -11.33, 95% CI [-20.99 to -1.66]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 3]; p = 0.1942, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -6.46, 95% CI [-16.23 to 3.30]

8. Secondary Outcome: Change in Fasting Plasma Glucose at Week 156
Description: Change in fasting plasma glucose (FPG) from baseline (week 0) to 156 weeks
Time Frame: week 0, week 156
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 230 | 234 | 242
mg/dL | -12.06 (3.8) | -5.45 (3.8) | 4.57 (3.62)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in fasting plasma glucose (FPG) from baseline to end of treatment at 156 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline FPG as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.0007, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -16.63, 95% CI [-26.19 to -7.06]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 8, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 2]; p = 0.0395, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -10.02, 95% CI [-19.56 to -0.49]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 8, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 3]; p = 0.1789, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -6.60, 95% CI [-16.24 to 3.03]

9. Secondary Outcome: Change in Mean Postprandial Glucose Based on Self-measured 8-point Plasma Glucose Profiles at Week 52
Description: Change in mean postprandial glucose (PPG) based on self-measured 8-point plasma glucose profiles from baseline (week 0) to 52 weeks (end of double-blind period). The 8 time points for self-measurements of plasma glucose were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner), at bedtime, and at 3:00 AM ± 30 min.
Time Frame: week 0, week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 191 | 187 | 182
mg/dL | -37.4 (3.37) | -30.8 (3.40) | -24.5 (3.32)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in mean postprandial glucose (PPG) from baseline to end of treatment at 52 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline PPG as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.0038, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -12.9, 95% CI [-21.6 to -4.2]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; Change in postprandial glucose (PPG) from baseline to end of treatment at 52 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline PPG as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 2]; p = 0.1616, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -6.3, 95% CI [-15.0 to 2.5]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 9, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 3]; p = 0.1319, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -6.6, 95% CI [-15.3 to 2.0]

10. Secondary Outcome: Change in Mean Postprandial Glucose Based on Self-measured 8-point Plasma Glucose Profiles at Week 104
Description: Change in mean postprandial glucose (PPG) based on self-measured 8-point plasma glucose profiles from baseline (week 0) to 104 weeks (end of 52-week extension). The 8 time points for self-measurements of plasma glucose were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner), at bedtime, and at 3:00 AM ± 30 min.
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 191 | 187 | 183
mg/dL | -37.15 (3.64) | -27.34 (3.68) | -24.85 (3.58)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in postprandial glucose (PPG) from baseline to end of treatment at 104 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline PPG as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.0105, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -12.30, 95% CI [-21.71 to -2.89]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 10, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 2]; p = 0.6060, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -2.49, 95% CI [-11.95 to 6.98]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 10, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 3]; p = 0.0392, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -9.81, 95% CI [-19.14 to -0.49]

11. Secondary Outcome: Change in Mean Postprandial Glucose Based on Self-measured 8-point Plasma Glucose Profiles at Week 156
Description: Change in mean postprandial glucose (PPG) based on self-measured 8-point plasma glucose profiles from baseline (week 0) to 156 weeks. The 8 time points for self-measurements of plasma glucose were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner), at bedtime, and at 3:00 AM ± 30 min.
Time Frame: week 0, week 156
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 191 | 187 | 183
mg/dL | -34.83 (3.65) | -25.68 (3.69) | -23.84 (3.59)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in postprandial glucose (PPG) from baseline to end of treatment at 156 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline PPG as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.0227, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -10.98, 95% CI [-20.42 to -1.54]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 11, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 2]; p = 0.7047, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -1.83, 95% CI [-11.33 to 7.66]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 11, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 3]; p = 0.0553, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -9.15, 95% CI [-18.51 to 0.21]

12. Primary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c) at Week 156
Description: Percentage point change in Glycosylated Haemoglobin A1c (HbA1c) from baseline (week 0) to 156 weeks
Time Frame: week 0, week 156
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage point of total HbA1c
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 234 | 236 | 241
percentage point of total HbA1c | -0.71 (0.09) | -0.44 (0.09) | -0.16 (0.08)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in glycosylated haemoglobin (HbA1c) from baseline to end of treatment at 156 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country, and previous oral antidiabetic drug (OAD) treatment as fixed effects and baseline HbA1c as covariate; Test type: Non-Inferiority or Equivalence — The two-sided 95% confidence interval (CI) for the treatment difference [liraglutide - glimepiride] was estimated. Liraglutide was shown to be non-inferior to glimepiride if the upper limit of the two-sided 95% CI for the treatment difference was below 0.4% and superior if the complete CI was below 0%; p < 0.0001, ANCOVA — The statistical analysis of the primary endpoint was done in a hierarchal manner due to multiple comparisons. No other adjustments were made for multiplicity. 2-sided significance level was 5%; Estimated treatment difference, LS Mean = -0.55, 95% CI [-0.77 to -0.34]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 12, analysis 1]; Test type: Non-Inferiority or Equivalence — The two-sided 95% confidence interval (CI) for the treatment difference [liraglutide - glimepiride] was estimated. Liraglutide was shown to be non-inferior to glimepiride if the upper limit of the two-sided 95% CI for the treatment difference was below 0.4% and superior if the complete CI was below 0%. Superiority of 1.2 mg liraglutide was only tested if 1.2 mg liraglutide was non-inferior to glimepiride and 1.8 mg liraglutide was superior to glimepiride; p = 0.0122, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Estimated treatment difference, LS Mean = -0.28, 95% CI [-0.49 to -0.06]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 12, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.0123, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -0.28, 95% CI [-0.49 to -0.06]

13. Secondary Outcome: Change in Prandial Increments of Plasma Glucose Based on Self-measured 8-point Plasma Glucose Profiles at Week 52
Description: Change in mean prandial increments of plasma glucose from baseline (week 0) to 52 weeks (end of double-blind period). The 8 time points for self-measured 8-point plasma glucose profiles were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner), at bedtime, and at 3:00 AM ± 30 min. Mean prandial increments of plasma glucose were calculated as the sum of the plasma glucose differences between post- and pre-meal values (for breakfast, lunch and dinner) divided by three.
Time Frame: week 0, week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 191 | 187 | 182
mg/dL | -9.6 (2.07) | -8.4 (2.10) | -5.6 (2.04)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in mean prandial increments of plasma glucose from baseline to end of treatment at 52 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.1396, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -4.0, 95% CI [-9.4 to 1.3]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 13, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 2]; p = 0.2968, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -2.9, 95% CI [-8.3 to 2.5]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; Change in postprandial (PPG) from baseline to end of treatment at 52 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 3]; p = 0.6639, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -1.2, 95% CI [-6.5 to 4.1]

14. Secondary Outcome: Change in Prandial Increments of Plasma Glucose Based on Self-measured 8-point Plasma Glucose Profiles at Week 104
Description: Change in mean prandial increments of plasma glucose from baseline (week 0) to 104 weeks (end of 52-week extension). The 8 time points for self-measured 8-point plasma glucose profiles were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner), at bedtime, and at 3:00 AM ± 30 min. Mean prandial increments of plasma glucose were calculated as the sum of the plasma glucose differences between post- and pre-meal values (for breakfast, lunch and dinner) divided by three.
Time Frame: week 0, week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 191 | 187 | 183
mg/dL | -11.76 (2.11) | -8.28 (2.14) | -7.95 (2.08)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in prandial increments of plasma glucose from baseline to end of treatment at 104 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.1720, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -3.81, 95% CI [-9.28 to 1.66]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 14, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 2]; p = 0.9060, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -0.33, 95% CI [-5.82 to 5.16]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 14, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 3]; p = 0.2089, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -3.48, 95% CI [-8.91 to 1.95]

15. Secondary Outcome: Change in Prandial Increments of Plasma Glucose Based on Self-measured 8-point Plasma Glucose Profiles at Week 156
Description: Change in mean prandial increments (incr.) of plasma glucose from baseline (week 0) to 156 weeks. The 8 time points for self-measured 8-point plasma glucose profiles were: before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner), at bedtime, and at 3:00 AM ± 30 min. Mean prandial increments of plasma glucose were calculated as the sum of the plasma glucose differences between post- and pre-meal values (for breakfast, lunch and dinner) divided by three.
Time Frame: week 0, week 156
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 191 | 187 | 183
mg/dL | -11.01 (2.11) | -7.53 (2.14) | -7.97 (2.07)
Statistical Analysis 1: Comparison: Lira 1.8 vs Glimepiride; Change in prandial increments of plasma glucose from baseline to end of treatment at 156 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment, country and previous anti-diabetic treatment as fixed effects and baseline value as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.2749, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -3.04, 95% CI [-8.51 to 2.42]
Statistical Analysis 2: Comparison: Lira 1.2 vs Glimepiride; [analysis description as in outcome 15, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 2]; p = 0.8765, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = 0.43, 95% CI [-5.05 to 5.92]
Statistical Analysis 3: Comparison: Lira 1.8 vs Lira 1.2; [analysis description as in outcome 15, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 3]; p = 0.2088, ANCOVA — 2-sided significance level 5%; Estimated treatment difference, LS Mean = -3.48, 95% CI [-8.90 to 1.95]

16. Secondary Outcome: Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes occuring from baseline (week 0) to 104 weeks (end of the 52-week extension). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 56 mg/dL. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 56 mg/dL.
Time Frame: weeks 0-104
Population: Full safety analysis set is all subjects who had been exposed to at least one dose of the study products.
Measure: Number; unit: episodes
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 246 | 251 | 248
episodes
  Major | 1 | 0 | 0
  Minor | 71 | 68 | 533
  Symptoms only | 87 | 133 | 405

17. Secondary Outcome: Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes occuring from week 104 to end of trial (week 195). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 56 mg/dL. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 56 mg/dL.
Time Frame: weeks 104-195
Population: Safety analysis set is all subjects who entered the year 3 extension at week 104.
Measure: Number; unit: episodes
Arm/Group | Lira 1.8 | Lira 1.2 | Glimepiride
Number analyzed (Participants) | 62 | 53 | 28
episodes
  Major | 0 | 0 | 1
  Minor | 13 | 3 | 34
  Symptoms only | 3 | 1 | 4

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time span of 195 weeks.
Description: The full safety analysis set is all subjects who had been exposed to at least one dose of the study products.
Groups:
- Lira 1.8 (Weeks 0-104): Liraglutide 1.8 mg once daily + glimepiride placebo 8 mg once daily, weeks 0-52 (double-blinded period) and open-label liraglutide 1.8 mg once daily in the extension period (weeks 52-104)
- Lira 1.2 (Weeks 0-104): Liraglutide 1.2 mg once daily + glimepiride placebo 8mg once daily, weeks 0-52 (double-blinded period) and open-label liraglutide 1.2 mg once daily in the extension period (weeks 52-104)
- Glimepiride (Weeks 0-104): Glimepiride 8 mg once daily + liraglutide placebo 200 mcl or liraglutide placebo 300 mcl, weeks 0-52 (double-blinded period) and open-label glimepiride 8 mg once daily in the extension period (weeks 52-104)
- Lira 1.8 (Weeks 104-195): Open-label liraglutide 1.8 mg once daily in the additional extension period (weeks 104-195)
- Lira 1.2 (Weeks 104-195): Open-label liraglutide 1.2 mg once daily in the additional extension period (weeks 104-195)
- Glimepiride (Weeks 104-195): Open-label glimepiride 8 mg once daily in the additional extension period (weeks 104-195)
Arm/Group | Lira 1.8 (Weeks 0-104) | Lira 1.2 (Weeks 0-104) | Glimepiride (Weeks 0-104) | Lira 1.8 (Weeks 104-195) | Lira 1.2 (Weeks 104-195) | Glimepiride (Weeks 104-195)
Serious Adverse Events (participants affected / at risk) | 22/246 | 23/251 | 20/248 | 5/62 | 1/53 | 2/28
Other Adverse Events (participants affected / at risk) | 183/246 | 181/251 | 148/248 | 40/62 | 37/53 | 13/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 1.8 (Weeks 0-104) (N=246) | Lira 1.2 (Weeks 0-104) (N=251) | Glimepiride (Weeks 0-104) (N=248) | Lira 1.8 (Weeks 104-195) (N=62) | Lira 1.2 (Weeks 104-195) (N=53) | Glimepiride (Weeks 104-195) (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenocortical Insufficiency Acute (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid Disorder (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis Perforated (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum Oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedematous Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess Limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridial Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic Coma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Grand Mal Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve Compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radial Nerve Palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral Stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 1.8 (Weeks 0-104) (N=246) | Lira 1.2 (Weeks 0-104) (N=251) | Glimepiride (Weeks 0-104) (N=248) | Lira 1.8 (Weeks 104-195) (N=62) | Lira 1.2 (Weeks 104-195) (N=53) | Glimepiride (Weeks 104-195) (N=28)
Nausea (Gastrointestinal disorders) | 75 (117) | 72 (97) | 21 (31) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 48 (66) | 44 (75) | 23 (37) | 5 (9) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 25 (36) | 33 (38) | 10 (12) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 29 (35) | 21 (24) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 13 (14) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 32 (42) | 36 (48) | 22 (30) | 8 (9) | 8 (10) | 1 (1)
Influenza (Infections and infestations) | 27 (37) | 23 (35) | 21 (27) | 3 (4) | 5 (8) | 2 (2)
Sinusitis (Infections and infestations) | 18 (31) | 21 (25) | 18 (24) | 4 (4) | 1 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 14 (18) | 26 (35) | 13 (15) | 6 (8) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 16 (21) | 23 (26) | 18 (19) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 9 (12) | 15 (17) | 11 (14) | 4 (4) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 18 (26) | 28 (53) | 23 (30) | 1 (2) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 19 (21) | 13 (19) | 13 (14) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (18) | 18 (21) | 17 (17) | 3 (3) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 11 (14) | 15 (15) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (15) | 9 (10) | 8 (9) | 1 (1) | 3 (3) | 0 (0)
Fatigue (General disorders) | 13 (15) | 8 (9) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 5 (6) | 11 (13) | 2 (2) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 14 (14) | 8 (11) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 11 (11) | 14 (14) | 17 (19) | 2 (2) | 6 (6) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 2 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial terminated due to an insufficient number of subjects remaining to obtain reasonable statistical power. Efficacy data was not analysed after week 156. Safety data was collected through week 195. No data was available from week 195 to 260

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones. This includes the right to not release interim results, because the release of such information can invalidate the results of the entire trial. At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.